# Effect of Immunoglobulin Plus Prednisolone in Reducing Coronary Artery Lesion in Patients with Kawasaki Disease

Trial Registration ID: NCT04078568

IRB Approval Date: 7 January, 2020

# Statistical Analysis Plan

The Data Management and Statistical Analysis Plan is directed to support the aims of the study

Version 3.0

July 30, 2020 Draft Oct 31, 2025 Modified

# Signed by:

| Fang Liu (Principal Investigator) | Fang Lin. |
|-----------------------------------|------------|
| Weili Yan (Senior Statistician) | WeiliYan |
| Yuanchen He (Statistician) | Yumchen He |

| SAP version history | | |
|---|---|---|
| Version Date | SAP Version | Details of Changes |
| July 30, 2020 | 1.1 | Draft |
| May 11, 2021 | 1.2 | Adding more secondary outcomes |
| May 19, 2023 | 1.3 | Adding more detail description of GEE model and secondary outcomes analyzation |
| June 15, 2023 | 1.4 | Adding solutions for non-convergence of GEE model |
| August 08, 2023 | 2.0 | Adjusting the structure of Introduction, as well as a few document styles and formats; adding more details about the definition of per-protocol population, primary outcome analyses and graphical displays. |
| October 31, 2025 | 3.0 | <ul> <li>Adding final solution for non-convergence of GEE model;</li> <li>Adding eight sensitivity analyses, with three of which suggested by reviewer;</li> <li>Adding post-hoc exploratory outcome analysis.</li> </ul> |

# Catalogue

| 1. | Introduction | 1 |
|---|---|---|
| 2. | Study Objective and Outcomes | 1 |
| | 2.1 Study Objective | 1 |
| | 2.2 Outcomes | 2 |
| | 2.2.1 Primary Outcome | 2 |
| | 2.2.2 Secondary Outcomes | 2 |
| | 2.2.3 Exploratory Outcomes | 4 |
| 3. | Study Design | 5 |
| | 3.1 Design. | 5 |
| | 3.2 Trial Sites | 5 |
| | 3.3 Interventions | 6 |
| | 3.3.1 Experimental arm: IVIG + Aspirin + Prednisolone | 6 |
| | 3.3.2 Control arm: Standard Treatment: IVIG + Aspirin | 7 |
| | 3.4 Randomization and Blinding. | 7 |
| | 3.5 Sample Size | 8 |
| 4. | Analysis Populations | 8 |
| | 4.1 Study Population Data Sets | 8 |
| | 4.2 Study Close Date | 9 |
| | 4.3 Data Monitoring and Cleaning | 9 |
| | 4.4 Data Check-up | . 10 |
| 5. | Statistical Analyses. | . 10 |
| | 5.1. Primary Outcome Analysis. | . 10 |
| | 5.1.1 ITT analysis of the primary outcome - the primary analysis | . 10 |
| | 5.1.2 Sensitivity analysis | . 11 |
| | 5.1.3 Subgroup analysis of the primary outcome | . 13 |
| | 5.2 Secondary Outcome Analysis | . 13 |
| | 5.2.1 Analysis of binary outcomes | . 14 |
| | 5.2.2 Analysis of continuous outcomes | . 14 |
| | 5.2.3 Analysis of time to event outcomes | . 15 |
| | 5.2.4 Analysis of other secondary outcomes (Exploratory Outcome Analysis) | |

| 5.3 Handling of Missing data | |
|---------------------------------------------|----|
| 6. General Considerations for Data Analyses | 16 |
| 6.1 Data Summaries | 16 |
| 6.2 Graphical Displays | 17 |
| 7. Study Variable List | 21 |
| 8. Reference | 38 |

### 1.Introduction

Kawasaki disease (KD), an acute systematic vasculitis, has been reported worldwide nowadays and more prevalent in Asia. Coronary artery lesion (CAL) is the most important complication and one of the main predictors to the long-term prognosis of KD. CAL can induce coronary artery aneurysm (CAA), occlusion, myocardial ischemia, myocardial infarction and even death, making KD a major cause of the acquired heart diseases in children. The large dose of intravenous immunoglobulin, together with aspirin (abbreviated as IVIG treatment) administered during the acute phase of KD has been well proved in reducing the occurrence of CALs. Given certain proportion of patients response poorly to this treatment, which is commonly linked with higher risk of CAL, it is worth exploring whether more aggressive treatments are able to achieve better effectiveness in reducing the incidence of CAL or not. Corticosteroid, preferred in the treatments of majority of vasculitis, remains controversial in the acute phase treatment of KD. Several studies suggest that the therapy time, regimen and the targeted people require careful considerations in the corticosteroid's treatment in KD. It is still under arguing that using corticosteroids in the initial treatment benefits all the KD patients rather than those with higher risk of IVIG resistance.

The purpose of this Statistical Analysis Plan (SAP) is to define the outcome variables, statistical methods and analysis strategies for a multicenter open-label randomized controlled trial. The trial aims to evaluate the effects of two therapies in reducing the incidence of CAL for children with acute KD: conventional IVIG treatment plus prednisolone (the experimental arm) and only IVIG treatment (the control arm).

# 2. Study Objective and Outcomes

### 2.1 Study Objective

This is a superiority randomized controlled trial, aiming to provide high quality evidence for

supporting effects and safety of current treatment combining steroid (corticosteroids) in the IVIG treatment plan for newly onset Kawasaki disease pediatric patients. The primary objective is to evaluate the hypothesis that IVIG treatment plus prednisolone will reduce the incidence of CAL at 1 month of illness comparing with the conventional IVIG treatment. The secondary objectives include comparing the need of additional treatment or not and duration of fever after initial treatment, occurrence of CAL after 1 month of illness onset, changes in laboratory data between two treatment groups, and serious adverse events.

### 2.2 Outcomes

### 2.2.1 Primary Outcome

The primary outcome is the occurrence of coronary artery lesions (CAL) at one month from disease onset. Two-dimensional echocardiography will be performed to evaluate CAL at six time points (at admission before treatment as the baseline, 2th week ( $\pm 2$  days), 1th month ( $\pm 5$  days), 3th month ( $\pm 5$  days), 6th month ( $\pm 5$  days), and 12th month ( $\pm 5$  days), respectively). The examination included the diameter of the left main coronary artery (LMCA), the left anterior descending artery (LAD), the left circumflex coronary artery (LCX), and the proximal and middle segments of the right coronary artery (RCA). Z scores of each coronary artery will be calculated<sup>1</sup>, and the occurrence of CAL is defined as  $z\geq 2$  of any coronary artery, including LMCA, LAD, LCX, and the proximal and middle segment of the RCA.

(Time Frame: at one month of illness) (Type: repeatedly measured binary variable)

### 2.2.2 Secondary Outcomes

1) Changes in z score of LMCA from admission. Data will be measured at six time points of illness: enrollment, 2th week (±2 days), 1th month (±5 days), 3th month (±5 days), 6th month (±5 days) and 12th month (±5 days), respectively.

(Time Frame: from admission to 12 months of illness) (Type: repeatedly measured continuous

variable)

- 2) Changes in z score of LAD from enrollment. Data will be measured at six time points of illness: enrollment, 2th week (±2 days), 1th month (±5 days), 3th month (±5 days), 6th month (±5 days) and 12th month (±5 days), respectively.
  - (Time Frame: from admission to 12 months of illness) (Type: repeatedly measured continuous variable)
- 3) Changes in z score of LCX from enrollment. Data will be measured at six time points of illness: enrollment, 2th week (±2 days), 1th month (±5 days), 3th month (±5 days), 6th month (±5 days) and 12th month (±5 days), respectively.
  - (Time Frame: from admission to 12 months of illness) (Type: repeatedly measured continuous variable)
- 4) Changes in z score of the proximal segment of RCA from enrollment. Data will be measured at six time points of illness: enrollment, 2th week (±2 days), 1th month (±5 days), 3th month (±5 days), 6th month (±5 days) and 12th month (±5 days), respectively.

  (Time Frame: from admission to 12 months of illness) (Type: repeatedly measured continuous
  - variable)
- 5) Changes in z score of the middle segment of RCA from enrollment. Data will be measured at six time points of illness: enrollment, 2th week (±2 days), 1th month (±5 days), 3th month (±5 days), 6th month (±5 days) and 12th month (±5 days), respectively.
  - (Time Frame: from admission to 12 months of illness) (Type: repeatedly measured continuous variable)
- 6) Need for additional treatment or not. The acute KD patients in both arms resistant to the initial IVIG therapy will be given additional treatment, which will be determined by the prescription record.
  - (Time Frame: at one month of illness) (Type: binary variable)
- 7) Duration (hours) of fever (defined as an axillary temperature <37.5 for more than 24 hours) after initiation of initial IVIG among participates of two arms.
  - (Time Frame: from initiation of initial IVIG infusion to the first record of being afebrile) (Type: time-to-event variable)
- 8) Change in serum C-reactive protein (CRP) concentration from admission to 72 hours after

completion of initial IVIG infusion.

(Time Frame: from admission to 72 hours after completion of initial IVIG infusion) (Type: continuous variable)

9) Serious adverse events (including death, hypertension, severe infection, allergic reactions, heart failure, thrombosis, etc.) will be recorded.

(Time Frame: from admission to 3 months of illness) (Type: character variable)

### 2.2.3 Exploratory Outcomes

The following exploratory outcomes were added by authors during manuscript drafting or suggested by reviewers during revision.

- 1) Occurrence of medium-to-giant CAAs. CAL classification was based on the maximum z score according to the 2017 American Heart Association guideline<sup>2</sup>. Medium CAA was defined as a maximum z score ≥5 to <10, and all internal diameters <8 mm; large or giant CAA was defined as a maximum z score ≥10, or any internal diameter ≥8 mm. Data were and will be collected at six time points of illness: enrollment, 2th week (±2 days), 1th month (±5 days), 3th month (±5 days), 6th month (±5 days) and 12th month (±5 days), respectively.
  - (Time Frame: from admission to 12 months of illness) (Type: repeatedly measured binary variable)
- 2) Occurrence of large/giant CAAs. Data were and will be collected at six time points of illness: enrollment, 2th week (±2 days), 1th month (±5 days), 3th month (±5 days), 6th month (±5 days) and 12th month (±5 days), respectively.
  - (Time Frame: from admission to 12 months of illness) (Type: binary variable)
- 3) Occurrence of CAL progression within 3 months of illness onset in all participants and those with CAL at baseline. CAL progression was defined as an increment in the z score ≥1 from baseline in any coronary artery (LMCA, LAD, LCX, proximal and middle segments of RCA) at any given time point within 3 months of illness onset.
  - (Time Frame: from admission to 3 months of illness) (Type: binary variable)
- 4) Changes in absolute diameters of LMCA, LAD, LCX, the proximal and middle segments of

RCA from enrollment. Data were and will be collected at six time points of illness: enrollment, 2th week (±2 days), 1th month (±5 days), 3th month (±5 days), 6th month (±5 days) and 12th month (±5 days), respectively.

(Time Frame: from admission to 12 months of illness) (Type: repeatedly measured continuous variable)

# 3. Study Design

### 3.1 Design

The trial is a multicenter, superiority, open-label, phase III randomized controlled trial. Patients fulfil the eligibility criteria as outlined in the protocol are invited to participate the trial consecutively and randomized individually to the control or experimental group. Randomization is based on the random block design (block size of 4).

### 3.2 Trial Sites

The trial will be conducted in 33 hospitals in China: Children's hospital of Fudan university, Jiangxi Provincial Children's Hospital, Qingdao Women and Children's Hospital, Chengdu Women's and Children's Central Hospital, Guangzhou Women and Children's Medical Center, Children's Hospital of Chongqing Medical University, Kaifeng Children's Hospital, Children's hospital of Soochow university, Xuzhou Children's Hospital, Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Shenzhen Children's Hospital, Shengjing Hospital of China Medical University, First Hospital of Jilin University, the third affiliated hospital of Zhengzhou university, Liuzhou Maternity and Children Healthcare Hospital, Inner Mongolia Autonomous Region People's Hospital, Hunan First People's Hospital, Henan Children's Hospital, Sichuan Academy of Medical Sciences & Sichuan Provincial People's Hospital, Children's Hospital of Nanjing Medical University, Union Hospital, Tongji Medical College, Huazhong University of

Science and Technology, Sun Yat-sen Memorial Hospital, Qilu Hospital of Shandong University, the First Affiliated Hospital of Zhengzhou University, Yuying Children's Hospital of Wenzhou Medical University, Xi'an Children's Hospital, Lanzhou University Second Hospital, Children's Hospital, Capital Institute of Pediatrics, Taihe Hospital Affiliated Hospital of Hubei University of Medicine, Anhui Children's Hospital, Shanghai Children's Hospital, and Bengbu First People's Hospital.

### 3.3 Interventions

### 3.3.1 Experimental arm: IVIG + Aspirin + Prednisolone

Patients in this arm will receive conventional IVIG treatment plus additional prednisolone 2 mg/kg per day in the initial treatment. The details are as follows:

In both arms, IVIG treatment is administered within 12 to 24 hours with the maximum dose of 60g. The dose of aspirin will be reduced to 3 to 5 mg/kg per day when fever subsides for 3 days and CRP is normal, and continued for at least 6 weeks after onset of KD. If patients resistant to initial IVIG therapy will be given rescue therapy, including a second dose of IVIG (2 g/kg), or a high dose of methylprednisolone (10 to 30 mg/kg per day), or infliximab (5 mg/kg), or other immunosuppressive agents, or a combination with two or more drugs, or even more aggressive treatment such as plasmapheresis, depending on patients' condition and physicians' experience. IVIG resistance is defined as recurrent or persistent fever (axillary temperature ≥37.5°C or rectal temperature ≥38°C) after 36 hours of completion of initial IVIG infusion.

Patients in the experimental group will additionally receive intravenous methylprednisolone 1.6 mg/kg per day which is given in 2 doses (equal to prednisolone 2 mg/kg, and the maximum dose is 60 mg of prednisolone), then switch to oral prednisolone 2 mg/kg when fever subsides for 3 days. If CRP returns to normal, the prednisolone dose will be tapered over 15 days in 5-day steps, from 2 mg/kg per day to 1 mg/kg per day then to 0.5 mg/kg per day. During corticosteroids administration, 0.5 mg/kg H2-blocker omeprazole will be given per day.

### 3.3.2 Control arm: Standard Treatment: IVIG + Aspirin

Patients in this arm will receive conventional treatment including, IVIG 2 g/kg and oral aspirin 30 mg/kg per day (given at 3 divided doses) in the initial treatment, which has been elaborated in the corresponding section of 3.3.1.

### 3.4 Randomization and Blinding

Randomization is stratified by trial sites and done in block size of 4. According to the random seeds, a sequence of study numbers and allocation plan will be generated by the SAS software (version 9.4). Each allocation sequence will be placed in four small, opaque and sealed envelopes numbered in order from 1 to 4, and then enclosed in a larger, opaque and sealed envelope marked with the block number. The randomized plan and concealed envelopes will be prepared by an independent statistician team from the Clinical Trial Unit (CTU) of the Children's Hospital of Fudan University, and delivered to and kept by the site coordinate nurse. Recruited patients will be randomly allocated in a 1:1 ratio to the control or experimental group based on the randomization plan. At each site, after obtaining signed informed consent from the eligible participant, the trained physician will meet with the prespecified institutional nurse to achieve the allocation plan as indicated by the corresponding envelope. The coordinate nurse will open the envelopes in numbered order according to the enrollment order, reveal the treatment allocation to the physician, and record the assignments of the enrolled patient.

Patients and physicians who treat patients will not be masked to the allocation, while pediatric cardiologists who assess CAL by echocardiography will be blinded to the allocation. All researchers conducting outcome assessments will be masked in the trial. The trial statistician will also be blinded regarding the treatment code when developing the statistical analysis plan and writing the statistical programs, which will be validated and completed using dummy randomization codes. The actual allocation will only be provided to the study team after lock of the database.

### 3.5 Sample Size

This study is a superiority trial. Sample size calculation is performed based on the difference of the primary outcome between the two arms. According to the previous study<sup>3</sup>, we assume a difference in the proportion of patients with CAL occurred within the first month of illness between the two groups of 3.3% (12.4% vs 9.1%, odds ratio [OR] = 0.73 for the control arm and the experimental arm, respectively). With an  $\alpha$  of 0.05 and a power of 0.8, a sample size of 1400 cases in each group will be needed. With an assumed dropout rate of 10%, a total of 3200 patients are planned for recruitment (1600 per arm).

# 4. Analysis Populations

### 4.1 Study Population Data Sets

Three study populations will be considered in the analysis. The primary analysis for the primary objective will be based on the intention-to-treatment population.

#### Intention-to-Treat population

Intention-to-treat (ITT) population will be defined at the moment the randomization is performed, including all subjects who are randomized.

Participants will be excluded from the ITT analysis if the primary outcome is missing, forming a modified ITT population (mITT).

#### Per-protocol population

Participants will be excluded from the per-protocol (PP) population if they:

- Being randomized but not receiving any treatment.

- Not adhering to allocated treatment due to:
  - aspirin allergy in either group.
  - being allocated to the experimental arm, while not completing the prednisolone treatment as recommended by the protocol (i.e., stopped early, took less than the recommended doses or tapered more quickly than the recommended period).
  - being allocated to the control arm but were prescribed additional prednisolone treatment due to discovered with IVIG resistance or other co-morbidities, such as juvenile idiopathic arthritis and necrotic lymphadenitis.

The treatment groups in the PP analysis will be determined according to what the participant actually received. This population will be used for the supportive analyses.

#### Safety population

Participants given any medicine-relate-treatments will be included in this population. Adverse reactions and events will be recorded. This population will be used for the safety analyses.

### **4.2 Study Close Date**

The data collection close date is the date on which the last patient completed 6-month follow-up.

All the participants will be followed up for 12 months.

### 4.3 Data Monitoring and Cleaning

Each center has a data manager dedicated to managing the data. Feedback on the inclusion of the week's study subjects is provided weekly in a WeChat group. All databases are synchronized in the cloud using NutCloud. The center data administrator verifies each sub-center database on a monthly basis. The data will then be checked to ensure that there are no erroneous entries and that all missing data is properly coded.

### 4.4 Data Check-up

Once all data have been inputted and checked, the database will be locked and a data download request made. The data will be downloaded into SAS, R and Stata formats for statistical analyses.

### 5. Statistical Analyses

### 5.1. Primary Outcome Analysis

# 5.1.1 ITT analysis of the primary outcome - the primary analysis

The primary analysis will be based on the ITT population as defined above. The primary outcome is a binary outcome: CAL occurs or not within 1 month of illness onset. Since CAL will be repeatedly examined at enrollment, 2 weeks, 1 month, 3 months, 6 months and 12 months respectively, generalized estimating equation (GEE) model will be performed, with treatment, visit and interaction between treatment with visit as fixed effect, patient ID as cluster effect, the mean of 5 coronary artery baseline z scores (described in section 2.2.1) as covariate variable. Risk difference (RD) and two-sided 95% confidence intervals (CI) between the two treatment groups will be estimated from the model using a binomial distribution and identity link function. OR with 95% CI at each time point will be obtained using GEE model with binomial distribution and logit link function. Binomial distribution and log link function will be used to obtain estimation of risk ratio (RR) and 95% CI. Exchangeable correlation structure is assumed for within-group variation for all the GEE models. The P value for the interaction term will be used to determine the statistical significance of the group difference at specific time point.

If the above GEE model does not converge, a poisson distribution will be used for the family function. A negative binomial distribution will be subsequently used for family function in case the GEE model based on poisson distribution does not converge. RD, OR and RR with their 95% CI

estimates will be reported by using identity, logit and log link function, respectively. In the final analysis, a normal family distribution was used because none of the three prespecified distribution models converged. RD and 95% CI estimates were derived using identity link function.

### 5.1.2 Sensitivity analysis

### 5.1.2.1 Per-protocol analysis of the primary outcome

A supportive analysis of the primary outcome will also be performed on the per-protocol population. Statistical methods will be the same as used in Section 5.1.1.

### 5.1.2.2 Covariate adjusted analysis of the primary outcome

An analysis of the primary endpoint will be adjusted for baseline information including age, body mass index (BMI), gender and complete or incomplete KD (following the KD diagnostic criteria from the American Heart Association released in 2017). From the above model, the adjusted estimates of RD and two-sided 95% CIs will be derived. The OR and RR with their 95% CIs will also be estimated from the GEE model using logit and log link function as described in Section 5.1.1.

Given the GEE model in the primary analysis has converged, if the GEE model doesn't converge when all covariates are introduced into the model simultaneously, the adjusted model will be established by removing a covariate one by one until the model converges.

### 5.1.2.3 Accounting for cluster effects of trial sites

A separate GEE model was applied to account for the cluster effects of trial sites, using the statistical method as described in Section 5.1.1. The RD with its 95% CI were estimated.

### 5.1.2.4 Best-case scenario

Participants with missing primary outcomes were assumed to have the best possible outcome, i.e., CAL did not occur at one month of illness onset in all of them. The statistical method was identical to that used in Section 5.1.1.

### 5.1.2.5 Worst-case scenario

Participants with missing primary outcomes were assumed to have the worst possible outcome, i.e., CAL occurred at one month of illness onset in all of them. The statistical method was identical to that used in Section 5.1.1.

### 5.1.2.6 Japanese criteria of CAL

The primary analysis (Section 5.1.1) was repeated using the Japanese Ministry of Health and Welfare criteria for CAL<sup>4</sup>, defined as follows:

- In children <5 years, any coronary artery diameter ≥3 mm; in children ≥5 years, ≥4 mm;
- Or  $\geq$ 1.5 times the diameter of an adjacent segment.

### 5.1.2.7 Z threshold $\geq$ 2.5 for CAL

The occurrence of CAL was re-defined as a z score ≥2.5 in any of the LMCA, LAD, LCX, or proximal/middle RCA segments. The same statistical method as in Section 5.1.1 was used.

### 5.1.2.8 CAL defined based on LAD and proximal RCA

The occurrence of CAL was re-defined as a z score ≥2 in either the LAD or proximal RCA segment.

The same statistical method as in Section 5.1.1 was used.

### 5.1.2.9 Adjusting for the baseline maximum z score

Using the same method as in Section 5.1.1, this sensitivity analysis adjusted for the maximum z score at baseline instead of the mean of 5 coronary artery baseline z scores.

### 5.1.2.10 GLM model analysis

This analysis used generalized linear model (GLM) treating response variable as a simple binary outcome without adjustment for any covariate. RD and 95% CI were estimated using a binomial distribution and an identity link function.

Sensitivity analyses 5.1.2.3 - 5.1.2.7 were conducted during manuscript preparation, and analyses 5.1.2.8 - 5.1.2.10 were added in response to reviewers' suggestions during manuscript revision.

### 5.1.3 Subgroup analysis of the primary outcome

Subgroup analyses will be performed for the primary outcome using GEE model as the primary analysis. We will stratify the analysis by age group (disease onset age <=1 or >1 year), gender (male or female), BMI group (according to different BMI distributions of age and gender in Chinese children, BMI will be stratified into three groups, underweight, normal weight, and overweight and obese, BMI percentile for age and gender of P10 and P85), complete or incomplete KD, IVIG respond or not and CAL presence or not at baseline. Same strategy and methods will be used as described in section 5.1.1.

Same strategy will be used when sensitivity analysis is performed for the secondary outcomes.

### **5.2 Secondary Outcome Analysis**

All secondary outcomes will be analyzed as for a superiority designed trial. Two-sided 95% CIs for

the treatment differences in these outcomes between two groups will be calculated and reported. Secondary outcome analyses will be based on the ITT population unless specified.

### 5.2.1 Analysis of binary outcomes

Repeated measured binary outcomes will be analyzed with the same tactics as that used for the primary outcome.

Non-repeated measured binary outcomes, referring to need for additional treatment or not, will be summarized by number (%) of participants by treatment group. The proportion difference will be tested by  $\chi^2$  methods or fisher exact test. If necessary for analysis, OR with their two-sided 95% CIs of the two groups will be derived from logistic regression. RR and 95% CI were also estimated using a binomial regression with log link function.

### 5.2.2 Analysis of continuous outcomes

The continuous outcome will be summarized using number of subjects (n), mean, standard deviation (SD), minimum, and maximum by intervention group. The repeated measured outcomes (including changes in z score of LMCA; changes in z score of LAD; changes in z score of LCX; changes in z score of the proximal segment of RCA; changes in z score of the middle segment of RCA) will be analyzed by generalized linear mixed model (GLMM) with intervention, visit and interaction between treatment with visit as fixed effect, patient ID as random effect, their baseline value as covariate variable. The outcomes which are not repeated measures (including change in serum C-reactive protein (CRP) concentration from admission to 72 hours after completion of initial IVIG infusion) will be analyzed by GLM. Gaussian distribution and identity link function will be used in the model. Difference in mean changes of outcome with their two-sided 95% confidence intervals between two groups will be estimated.

### 5.2.3 Analysis of time to event outcomes

Kaplan-Meier method will be used to plot cumulative event rate of time to first event data. If the Kaplan-Meier curves don't cross, log-rank test will be performed to detect a difference between groups. Cox regression will be performed when the proportional hazards assumption is met and hazard ratio and 95% CI will be estimated.

If the Kaplan-Meier curves cross or the proportional hazards assumption is not satisfied, the win ratio method<sup>5</sup> will be performed.

# 5.2.4 Analysis of other secondary outcomes (Exploratory Outcome Analysis)

The post-hoc secondary outcomes were analyzed using the same statistical methods described above unless otherwise specified. Specifically, these exploratory outcomes included: occurrence of medium-to-giant CAAs among all participants (Section 5.2.1, repeated measured binary outcomes); CAL progression among all participants (Section 5.2.1, non-repeated measured binary outcomes); and changes in absolute diameters of LMCA, LAD, LCX, the proximal and middle segments of RCA (Section 5.2.2, repeated measured continuous outcomes).

Considering the low incidence of large/giant CAAs (<1%), between-group RRs and two-sided 95% CIs were estimated from a GLM with a negative binomial distribution and log link, adjusting for the mean baseline z scores. Participants with large/giant aneurysms at baseline were excluded from this analysis.

For analysis of CAL progression in participants with baseline CAL, the model was further adjusted for age, sex, KD type, baseline sodium level, CRP concentration, and white blood cell count. RR and corresponding 95% CI were estimated.

### 5.3 Handling of Missing data

Missing baseline covariates will be imputed using simple imputation methods in the covariate adjusted analysis based on the covariate distributions, should the missing values for a particular covariate be less than 5%. For a continuous variable, missing values will be imputed from random values from a permutated normal distribution with mean and SD calculated from the available sample. For a categorical variable, missing values will be imputed from random values from a uniform distribution with probabilities P1, P2, ..., and Pk from the sample. The seed to be used is 20230605. We do not assume the condition that missing of covariate variable at baseline will be over 5%.

# 6. General Considerations for Data Analyses

SAS (version 9.4) will be used to perform all data analyses and generate majority of data displays. STATA® (version 16.0) or R may also be used for some data analyses and generating statistical graphs. All analyses for the primary and secondary outcome variables will be primarily based on ITT population. Two-side tests and P values will be reported. Regression models for repeated measurement will be used for outcomes that are repeatedly measured, group differences at the prespecified timepoint will be computed and reported.

### 6.1 Data Summaries

Continuous variables will be summarized according to number of subjects with non-missing data (n), mean, standard deviation (SD), median, minimum, maximum and range interquartile (IQR). The confidence intervals will be reported on summaries of continuous effectiveness variables. Categorical variables will be summarized according to the absolute frequency and percentage of subjects (%) in each category level. The denominator for the percentages is the number of subjects in the treatment arm with data available, unless noted otherwise.

# **6.2** Graphical Displays

Table 1. Baseline characteristics of patients

Analysis Set: ITT population

| Statistic (N=) (N=) (N=) | | Anarysi | is Set: ITT popul | | |
|---|---|---|---|---|---|
| Gender, n (%) Female Male Male Age (years) n Mean (SD) Median (IQR) Min-Max Height (cm) Mean (SD) Median (IQR) Min-Max Weight (kg) Mean (SD) Median (IQR) Min-Max Min-Max LMCA n Median (IQR) Median (IQR) Min-Max LAD Mean (SD) Median (IQR) Mean (SD) Median (IQR) Mean (SD) Median (IQR) Min-Max LCX LCX n | Variable | Statistic | Treatment A | Treatment B | All |
| Age (years) n Mean (SD) Median (IQR) Min-Max Min-Max Height (cm) n Median (IQR) Median (IQR) Min-Max Median (IQR) Weight (kg) n Median (IQR) Min-Max LMCA n Mean (SD) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Mean (SD) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Min-Max Median (IQR) Min-Max Min-Max LCX n | | | (IN=) | (IN=) | (IN=) |
| Age (years) n Mean (SD) Median (IQR) Min-Max Height (cm) Mean (SD) Median (IQR) Min-Max Weight (kg) Mean (SD) Median (IQR) Min-Max Min-Max LMCA n Mean (SD) Median (IQR) Median (IQR) Min-Max LAD n Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Min-Max Min-Max LCX n | Gender, n (%) | Female | | | |
| Mean (SD) Median (IQR) Min-Max Height (cm) Mean (SD) Median (IQR) Min-Max Weight (kg) Median (IQR) Median (IQR) Min-Max Median (IQR) Median (IQR) Median (IQR) Mean (SD) Median (IQR) Min-Max LAD Mean (SD) Median (IQR) Min-Max LCX Mean (SD) Mean (SD) | | Male | | | |
| Median (IQR) Min-Max Height (cm) n Mean (SD) Median (IQR) Min-Max Weight (kg) n Median (IQR) Min-Max LMCA n Mean (SD) Median (IQR) Min-Max LAD n Mean (SD) Median (IQR) Min-Max LCX n Mean (SD) | Age (years) | n | | | |
| Min-Max | | Mean (SD) | | | |
| Height (cm) n Mean (SD) Median (IQR) Min-Max Weight (kg) n Mean (SD) Median (IQR) Min-Max LMCA n Mean (SD) Median (IQR) Min-Max LAD n Mean (SD) Mean (SD) Mean (SD) Mean (SD) Min-Max LAD n Mean (SD) Median (IQR) Min-Max LAD Mean (SD) | | Median (IQR) | | | |
| Mean (SD) Median (IQR) Min-Max Min-Max Weight (kg) n Mean (SD) Median (IQR) Min-Max LMCA Mean (SD) Median (IQR) Min-Max LAD Mean (SD) Median (IQR) Median (IQR) Min-Max LAD Median (IQR) Median (IQR) Min-Max LCX n Mean (SD) Mean (SD) | | Min-Max | | | |
| Median (IQR) Min-Max Weight (kg) n Mean (SD) Median (IQR) Min-Max LMCA n Mean (SD) Median (IQR) Median (IQR) Min-Max LAD n Mean (SD) Median (IQR) Min-Max LAD n Mean (SD) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Median (IQR) Min-Max LCX n Mean (SD) | Height (cm) | n | | | |
| Weight (kg) n Mean (SD) Median (IQR) Min-Max Min-Max LMCA n Mean (SD) Median (IQR) Min-Max Min-Max LAD n Median (SD) Median (IQR) Min-Max Min-Max LCX n Mean (SD) Mean (SD) | | Mean (SD) | | | |
| Weight (kg) n Mean (SD) Median (IQR) Min-Max Min-Max LMCA n Mean (SD) Median (IQR) Min-Max Min-Max LAD n Mean (SD) Median (IQR) Median (IQR) Min-Max LCX n Mean (SD) Mean (SD) | | Median (IQR) | | | |
| Mean (SD) Median (IQR) Min-Max LMCA n Mean (SD) Median (IQR) Min-Max LAD n Mean (SD) Median (IQR) Min-Max LCX n Mean (SD) | | Min-Max | | | |
| Median (IQR) | Weight (kg) | n | | | |
| Min-Max | | Mean (SD) | | | |
| LMCA n Mean (SD) Median (IQR) Min-Max Min-Max LAD n Mean (SD) Median (IQR) Min-Max Min-Max LCX n Mean (SD) Mean (SD) | | Median (IQR) | | | |
| Mean (SD) | | Min-Max | | | |
| Median (IQR) | LMCA | n | | | |
| Min-Max | | Mean (SD) | | | |
| LAD n Mean (SD) Median (IQR) Min-Max LCX Mean (SD) Mean (SD) | | Median (IQR) | | | |
| Mean (SD) Median (IQR) Min-Max LCX n Mean (SD) | | Min-Max | | | |
| Median (IQR) Min-Max LCX n Mean (SD) | LAD | n | | | |
| LCX n Mean (SD) | | Mean (SD) | | | |
| LCX n Mean (SD) | | Median (IQR) | | | |
| Mean (SD) | | Min-Max | | | |
| | LCX | n | | | |
| Median (IOR) | | Mean (SD) | | | |
| iviculaii (iQiC) | | Median (IQR) | | | |

| Variable | Statistic | Treatment A (N=) | Treatment B (N=) | All (N=) |
|------------|--------------|------------------|------------------|----------|
| | Min-Max | | | |
| RCA (prox) | n | | | |
| | Mean (SD) | | | |
| | Median (IQR) | | | |
| | Min-Max | | | |
| RCA (mid) | n | | | |
| | Mean (SD) | | | |
| | Median (IQR) | | | |
| | Min-Max | | | |

Table 2. Summary for primary outcomes by generalized estimating equation model

Analysis Set: ITT population

| | | Participants, No. (%) | | Generalized estimating equation model analysis | | |
|---|---|---|---|---|---|---|
| Primary outcome | Visit | Treatment A | Treatment B | Risk difference | Odds Ratio | Risk ratio |
| | | | | (95% CI) | (95% CI) | (95% CI) |
| Covariate unadjusted | a | | | T | | |
| CAL | 1 month | | | | | |
| | 3 months | | | | | |
| | 6 months | | | | | |
| | 12 months | | | | | |
| Covariate adjusted <sup>b</sup> | | | | | | |
| CAL | 1 month | | | | | |
| | 3 months | | | | | |
| | 6 months | | | | | |
| | 12 months | | | | | |

<sup>&</sup>lt;sup>a</sup>The GEE model only includes the mean of 5 coronary artery baseline z scores as covariate.

Table 3. Subgroup analysis of primary outcome by generalized estimating equation model

<sup>&</sup>lt;sup>b</sup>The GEE model was adjusted by including ...as covariates.

### Analysis Set: ITT population

| | | | Participan | ts, No. (%) | Generalized est | imating equation | model analysis |
|---|---|---|---|---|---|---|---|
| Primary outcome | Variable | Visit | Treatment A | Treatment B | Risk difference (95%CI) | Odds ratio<br>(95%CI) | Risk ratio (95%CI) |
| CAL | Age (<=1 year) | 1 month | | | | | |
| | | 3 months | | | | | |
| | | 6 months | | | | | |
| | | 12 months | | | | | |
| | Age (>1 year) | 1 month | | | | | |
| | | 3 months | | | | | |
| | | 6 months | | | | | |
| | | 12 months | | | | | |
| | Gender (F) | 1 month | | | | | |
| | | 3 months | | | | | |
| | | 6 months | | | | | |
| | | 12 months | | | | | |
| | Gender (M) | 1 month | | | | | |
| | | 3 months | | | | | |
| | | 6 months | | | | | |
| | | 12 months | | | | | |
| | BMI (l) | 1 month | | | | | |
| | | 3 months | | | | | |
| | | 6 months | | | | | |
| | | 12 months | | | | | |
| | BMI (N) | 1 month | | | | | |
| | | 3 months | | | | | |
| | | 6 months | | | | | |
| | | 12 months | | | | | |
| | BMI (H) | 1 month | | | | | |
| | | 3 months | | | | | |
| | | 6 months | | | | | |

| | | | Participants, No. (%) | | Generalized estimating equation model analysis | | |
|---|---|---|---|---|---|---|---|
| Primary outcome | Variable | Visit | Treatment A | Treatment B | Risk difference (95%CI) | Odds ratio<br>(95%CI) | Risk ratio (95%CI) |
| | | 12 months | | | | | |

Table 4. Secondary analysis by generalized estimating equation model Analysis Set: ITT population

| | | n, mea | un (SD) | Generalized estimating equation model analysis | |
|---|---|---|---|---|---|
| Secondary outcome | Visit | Treatment A (N=) | Treatment B (N=) | Risk difference (95% CI) | P value |
| LMCA | 1 month | | | | |
| | 3 months | | | | |
| | 6 months | | | | |
| | 12 months | | | | |
| LAD | 1 month | | | | |
| | 3 months | | | | |
| | 6 months | | | | |
| | 12 months | | | | |
| LCX | 1 month | | | | |
| | 3 months | | | | |
| | 6 months | | | | |
| | 12 months | | | | |
| RCA (prox) | 1 month | | | | |
| | 3 months | | | | |
| | 6 months | | | | |
| | 12 months | | | | |
| RCA (mid) | 1 month | | | | |
| | 3 months | | | | |
| | 6 months | | | | |
| | 12 months | | | | |

# 7. Study Variable List

Table 1 Variable list

Note: T, text variable; D, The date type; N, Continuous variable; B, binary variable; C, categorical variable

| No | Variable | Variable Type | Variable interpretation |
|---|---|---|---|
| 1 | center | Т | Name of center |
| 2 | id_center | Т | Number of center |
| 3 | name_pat | Т | Acronym of subject |
| 4 | patid | N | Study ID of subject |
| 5 | time_start | D | Date of enrollment |
| 6 | time_end | D | Date of end |
| 7 | investigator | | Investigator signature |
| 8 | inc_1 | В | Meeting the diagnostic criteria of |
| | | | Kawasaki disease |
| 9 | inc_2 | В | Age≥1 month and weight≤30kg |
| 10 | inc_3 | В | Fever≤10 days |
| 11 | inc_4 | В | All coronary z values are <10 before IVIG |
| | | | administration |
| 12 | inc_5 | В | Able to complete follow-up |
| 13 | inc_6 | В | The guardian is fully informed and signs the |
| | | | informed consent |
| 14 | exclusion_1 | В | Use of hormones or other |
| | | | immunosuppressants 1 month before KD |
| | | | onset |
| 15 | exclusion_2 | В | Recurrence of KD |

| 16 | exclusion_3 | В | Body temperature is normal at the time of |
|---|---|---|---|
| | | | inclusion (T≤37.5≥24h) |
| 17 | exclusion_4 | В | With the following infections: sepsis, septic |
| | | | meningitis, peritonitis, bacterial pneumonia, |
| | | | varicella, and influenza |
| 18 | exclusion_5 | В | History of serious immune diseases, such as |
| | | | immunodeficiency, or chromosomal |
| | | | abnormalities |
| 19 | eligibility | В | Eligibility or not |
| 20 | arm | Т | Intervention allocation |
| 21 | gender | В | Gender |
| 22 | birth | D | Date of birth |
| 23 | tel | Т | Telephone |
| 24 | height | N | Height at baseline |
| 25 | weight | N | Body weight at baseline |
| 26 | id_hospital | Т | Hospital admission number |
| 27 | date_fisrt_fever | D | Date of first fever |
| 28 | date_ivig_on | D | Start date of IVIG administration |
| 29 | hour_ivig_on | N | Start time of IVIG administration |
| 30 | manifes_fever | В | Clinical feature - fever |
| 31 | manifes_fever_days | N | Clinical feature - febrile days |
| 32 | manifes_fever_high | N | Clinical feature - maximum heating |
| | | | temperature |
| 33 | manifes_conjestion | В | Clinical feature - conjunctivitis |
| 34 | manifes_rash | В | Clinical feature - rash |
| 35 | manifes_tongue | В | Clinical feature - oral changes |
| 36 | manifes_swollen_hand | В | Clinical feature - extremity changes |
| 37 | manifes_lymph | В | Clinical feature - cervical lymphadenopathy |
| 38 | manifes_crissum | В | Clinical feature - perianal vulva flushing and |

| | | | molting |
|----|-----------------|---|--------------------------------------------|
| 39 | maniffes_scar | В | Clinical feature - red and swollen kaba |
| 40 | manifes_oth | В | Clinical feature - other |
| 41 | manifes_oth_txt | Т | Clinical feature - other text |
| 42 | a_tempstart | N | Body temperature at IVIG administration |
| | | | begin |
| 43 | a_notestart | Т | Note of body temperature at IVIG |
| | | | administration begin |
| 44 | a_temp0h | N | Body temperature at IVIG administration |
| | | | end |
| 45 | a_note0h | Т | Note of body temperature at IVIG |
| | | | administration end |
| 46 | a_temp6h | N | Body temperature at 6 hours after IVIG |
| | | | administration |
| 47 | a_note6h | Т | Note of body temperature at 6 hours after |
| | | | IVIG administration |
| 48 | a_temp12h | N | Body temperature at 12 hours after IVIG |
| | | | administration |
| 49 | a_note12h | Т | Note of body temperature at 12 hours after |
| | | | IVIG administration |
| 50 | a_temp18h | N | Body temperature at 18 hours after IVIG |
| | | | administration |
| 51 | a_note18h | Т | Note of body temperature at 18 hours after |
| | | | IVIG administration |
| 52 | a_temp24h | N | Body temperature at 24 hours after IVIG |
| | | | administration |
| 53 | a_note24h | Т | Note of body temperature at 24 hours after |
| | | | IVIG administration |
| 54 | a_temp30h | N | Body temperature at 30 hours after IVIG |

| | | | administration |
|----|-----------|---|----------------------------------------------|
| 55 | a_note30h | Т | Note of body temperature at 30 hours after |
| | | | IVIG administration |
| 56 | a_temp36h | N | Body temperature at 36 hours after IVIG |
| | | | administration |
| 57 | a_note36h | Т | Note of body temperature at 36 hours after |
| | | | IVIG administration |
| 58 | a_temp42h | N | Body temperature at 42 hours after IVIG |
| | | | administration |
| 59 | a_note42h | Т | Note of body temperature at 42 hours after |
| | | | IVIG administration |
| 60 | a_temp48h | N | Body temperature at 48 hours after IVIG |
| | | | administration |
| 61 | a_note48h | Т | Note of body temperature at 48 hours after |
| | | | IVIG administration |
| 62 | a_temp54h | N | Body temperature at 54 hours after IVIG |
| | | | administration |
| 63 | a_note54h | Т | Note of body temperature at 54 hours after |
| | | | IVIG administration |
| 64 | a_temp60h | N | Body temperature at 60 hours after IVIG |
| | | | administration |
| 65 | a_note60h | Т | Note of body temperature at 60 hours after |
| | | | IVIG administration |
| 66 | b1_wbc0 | N | White blood cell counts before IVIG |
| | | | administration |
| 67 | b1_wbc3d | N | White blood cell counts at 72 hours after |
| | | | IVIG administration |
| 68 | b1_wbc6d | N | White blood cell counts at 6 days after IVIG |
| | | | administration |

| 69 | b1_wbc9d | N | White blood cell counts at 9 days after IVIG |
|----|----------------|---|----------------------------------------------|
| | | | administration |
| 70 | b2_neutro0 | N | Neutrophil counts before IVIG |
| | | | administration |
| 71 | b2_neutro3d | N | Neutrophil counts at 72 hours after IVIG |
| | | | administration |
| 72 | b2_neutro6d | N | Neutrophil counts at 6 days after IVIG |
| | | | administration |
| 73 | b2_neutro9d | N | Neutrophil counts at 9 days after IVIG |
| | | | administration |
| 74 | b3_platelet0 | N | Blood platelet before IVIG administration |
| 75 | b3_platelet3d | N | Blood platelet at 72 hours after IVIG |
| | | | administration |
| 76 | b3_platelet6d | N | Blood platelet at 6 days after IVIG |
| | | | administration |
| 77 | b3_platelet9d | N | Blood platelet at 9 days after IVIG |
| | | | administration |
| 78 | b4_hemoglob10 | N | Hemoglobin before IVIG administration - 1 |
| 79 | b4_hemoglob20 | N | Hemoglobin before IVIG administration - 2 |
| 80 | b4_hemoglob13d | N | Hemoglobin at 72 hours after IVIG |
| | | | administration - 1 |
| 81 | b4_hemoglob23d | N | Hemoglobin at 72 hours after IVIG |
| | | | administration - 2 |
| 82 | b4_hemoglob16d | N | Hemoglobin at 6 days after IVIG |
| L | | | administration - 1 |
| 83 | b4_hemoglob26d | N | Hemoglobin at 6 days after IVIG |
| | | | administration - 2 |
| 84 | b4_hemoglob19d | N | Hemoglobin at 9 days after IVIG |
| | | | administration - 1 |

| 85 | b4_hemoglob29d | N | Hemoglobin at 9 days after IVIG |
|-----|-----------------|---|---------------------------------------------|
| | | | administration - 2 |
| 86 | b4_hemoglobunit | Т | Unit of hemoglobin |
| 87 | b5_hct0 | N | HCT before IVIG administration |
| 88 | b5_hct3d | N | HCT at 72 hours after IVIG administration |
| 89 | b5_hct6d | N | HCT at 6 days after IVIG administration |
| 90 | b5_hct9d | N | HCT at 9 days after IVIG administration |
| 91 | b6_crp10 | N | CRP before IVIG administration - 1 |
| 92 | b6_crp20 | N | CRP before IVIG administration - 2 |
| 93 | b6_crp13d | N | CRP at 72 hours after IVIG administration - |
| | | | 1 |
| 94 | b6_crp23d | N | CRP at 72 hours after IVIG administration - |
| | | | 2 |
| 95 | b6_crp16d | N | CRP at 6 days after IVIG administration - 1 |
| 96 | b6_crp26d | N | CRP at 6 days after IVIG administration - 2 |
| 97 | b6_crp19d | N | CRP at 9 days after IVIG administration -1 |
| 98 | b6_crp29d | N | CRP at 9 days after IVIG administration - 2 |
| 99 | b6_crpunit | Т | Unit of CRP |
| 100 | b7_saa0 | N | Serum amyloid A before IVIG |
| | | | administration |
| 101 | b7_saa3d | N | Serum amyloid A at 72 hours after IVIG |
| | | | administration |
| 102 | b7_saa6d | N | Serum amyloid A at 6 days after IVIG |
| | | | administration |
| 103 | b7_saa9d | N | Serum amyloid A at 9 days after IVIG |
| | | | administration |
| 104 | c1_esr0 | N | Erythrocyte sedimentation rate (ESR) |
| | | | before IVIG administration |
| | c1 esr4 | N | Erythrocyte sedimentation rate (ESR) after |

| | | | IVIG administration |
|-----|---------------|---|-------------------------------------------|
| 106 | c2_alb0 | N | Albumin before IVIG administration |
| 107 | c2_alb4 | N | Albumin after IVIG administration |
| 108 | c3_prealb10 | N | Prealbumin before IVIG administration - 1 |
| 109 | c3_prealb14 | N | Prealbumin after IVIG administration - 1 |
| 110 | c3_prealb20 | N | Prealbumin before IVIG administration - 2 |
| 111 | c3_prealb24 | N | Prealbumin after IVIG administration - 2 |
| 112 | c3_prealb30 | N | Prealbumin before IVIG administration - 3 |
| 113 | c3_prealb34 | N | Prealbumin after IVIG administration - 3 |
| 114 | c3_prealbunit | Т | Unit of prealbumin |
| 115 | c4_gpt10 | N | Glutamic-pyruvic transaminase before |
| | | | IVIG administration - 1 |
| 116 | c4_gpt14 | N | Glutamic-pyruvic transaminase after IVIG |
| | | | administration - 1 |
| 117 | c4_gpt20 | N | Glutamic-pyruvic transaminase before |
| | | | IVIG administration - 2 |
| 118 | c4_gpt24 | N | Glutamic-pyruvic transaminase after IVIG |
| | | | administration - 2 |
| 119 | c4_gptunit | Т | Unit of glutamic-pyruvic transaminase |
| 120 | c5_got10 | N | Glutamic oxalacetic transaminase before |
| | | | IVIG administration - 1 |
| 121 | c5_got14 | N | Glutamic oxalacetic transaminase after |
| | | | IVIG administration - 1 |
| 122 | c5_got20 | N | Glutamic oxalacetic transaminase before |
| | | | IVIG administration - 2 |
| 123 | c5_got24 | N | Glutamic oxalacetic transaminase after |
| | | | IVIG administration - 2 |
| 124 | c5_gotunit | Т | Unit of glutamic oxalacetic transaminase |
| | | 1 | |

| | | | 1 |
|-----|----------------|---|---------------------------------------------|
| 126 | c6_glucose14 | N | Blood glucose after IVIG administration - 1 |
| 127 | c6_glucose20 | N | Blood glucose before IVIG administration - |
| | | | 2 |
| 128 | c6_glucose24 | N | Blood glucose after IVIG administration - 2 |
| 129 | c6_glucoseunit | Т | Unit of blood glucose |
| 130 | c7_ckmb10 | N | Creatine kinase isoenzyme before IVIG |
| | | | administration - 1 |
| 131 | c7_ckmb14 | N | Creatine kinase isoenzyme after IVIG |
| | | | administration - 1 |
| 132 | c7_ckmb20 | N | Creatine kinase isoenzyme before IVIG |
| | | | administration - 2 |
| 133 | c7_ckmb24 | N | Creatine kinase isoenzyme after IVIG |
| | | | administration - 2 |
| 134 | c7_ckmb30 | N | Creatine kinase isoenzyme before IVIG |
| | | | administration - 3 |
| 135 | c7_ckmb34 | N | Creatine kinase isoenzyme after IVIG |
| | | | administration - 3 |
| 136 | c7_ckmunit | Т | Unit of creatine kinase isoenzyme |
| 137 | c8_bnp0 | N | B-type natriuretic peptide before IVIG |
| | | | administration |
| 138 | c8_bnp4 | N | B-type natriuretic peptide after IVIG |
| | | | administration |
| 139 | c9_probnp10 | N | N-terminal moiety of B-type natriuretic |
| | | | peptide before IVIG administration - 1 |
| 140 | c9_probnp14 | N | N-terminal moiety of B-type natriuretic |
| | | | peptide after IVIG administration - 1 |
| 141 | c9_probnp20 | N | N-terminal moiety of B-type natriuretic |
| | | | peptide before IVIG administration - 2 |

| 142 | c9_probnp24 | N | N-terminal moiety of B-type natriuretic |
|-----|------------------|---|--------------------------------------------|
| | | | peptide after IVIG administration - 2 |
| 143 | c9_probnpunit | Т | Unit of N-terminal moiety of B-type |
| | | | natriuretic peptide |
| 144 | c10_sodium0 | N | Sodium before IVIG administration |
| 145 | c10_sodium4 | N | Sodium after IVIG administration |
| 146 | c11_troponin10 | N | Serum troponin before IVIG administration |
| | | | - 1 |
| 147 | c11_troponin14 | N | Serum troponin after IVIG administration - |
| | | | 1 |
| 148 | c11_troponin20 | N | Serum troponin before IVIG administration |
| | | | - 2 |
| 149 | c11_troponin24 | N | Serum troponin after IVIG administration - |
| | | | 2 |
| 150 | c11_troponin30 | N | Serum troponin before IVIG administration |
| | | | - 3 |
| 151 | c11_troponin34 | N | Serum troponin after IVIG administration - |
| | | | 3 |
| 152 | c11_troponin40 | N | Serum troponin before IVIG administration |
| | | | - 4 |
| 153 | c11_troponin44 | N | Serum troponin after IVIG administration - |
| | | | 4 |
| 154 | c11_troponinunit | Т | Unit of serum troponin |
| 155 | c12_tspot0 | N | T-SPOT before IVIG administration |
| 156 | c12_tspot4 | N | T-SPOT after IVIG administration |
| 157 | c13_tbil0 | N | Serum total bilirubin before IVIG |
| | | | administration |
| 158 | c13_tbil4 | N | Serum total bilirubin after IVIG |
| | | | administration |

| | T | 1 | T |
|-----|-------------|---|---------------------------------------------|
| 159 | c14_tg10 | N | Triglyceride before IVIG administration - 1 |
| 160 | c14_tg14 | N | Triglyceride after IVIG administration - 1 |
| 161 | c14_tg20 | N | Triglyceride before IVIG administration - 2 |
| 162 | c14_tg24 | N | Triglyceride after IVIG administration - 1 |
| 163 | c14_tgunit | Т | Unit of Triglyceride |
| 164 | c15_tc10 | N | Total cholesterol before IVIG |
| | | | administration - 1 |
| 165 | c15_tc14 | N | Total cholesterol after IVIG administration |
| | | | - 1 |
| 166 | c15_tc20 | N | Total cholesterol before IVIG |
| | | | administration - 2 |
| 167 | c15_tc24 | N | Total cholesterol after IVIG administration |
| | | | - 2 |
| 168 | c15_tcunit | Т | Unit of total cholesterol |
| 169 | c16_ldl10 | N | LDL before IVIG administration - 1 |
| 170 | c16_ldl14 | N | LDL after IVIG administration - 1 |
| 171 | c16_ldl20 | N | LDL before IVIG administration - 2 |
| 172 | c16_ldl24 | N | LDL after IVIG administration - 2 |
| 173 | c16_ldlunit | Т | Unit of LDL |
| 174 | c17_dimer10 | N | D-dimer before IVIG administration - 1 |
| 175 | c17_dimer14 | N | D-dimer after IVIG administration - 1 |
| 176 | c17_dimer20 | N | D-dimer before IVIG administration - 2 |
| 177 | c17_dimer24 | N | D-dimer after IVIG administration - 2 |
| 178 | c17_dimer30 | N | D-dimer before IVIG administration - 3 |
| 179 | c17_dimer34 | N | D-dimer after IVIG administration - 3 |
| 180 | c17_dimer40 | N | D-dimer before IVIG administration - 4 |
| 181 | c17_dimer44 | N | D-dimer after IVIG administration - 4 |
| 182 | c17_dimer50 | N | D-dimer before IVIG administration - 5 |
| 183 | c17_dimer54 | N | D-dimer after IVIG administration - 5 |
| | | • | |

| 184 | c17_dimerunit | Т | Unit of D-dimer |
|---|---|---|---|
| 185 | c18_pct0 | N | Calcitonin before IVIG administration |
| 186 | c18_pct4 | N | Calcitonin after IVIG administration |
| 187 | c19_il60 | N | IL-6 before IVIG administration |
| 188 | c19_il64 | N | IL-6 after IVIG administration |
| 189 | c20_tnf0 | N | TNF before IVIG administration |
| 190 | c20_tnf4 | N | TNF after IVIG administration |
| 191 | d1_date_ucg0 | D | Date of ultrasonic cardiogram before IVIG administration |
| 192 | d1_date_ucg5 | D | Date of ultrasonic cardiogram at 2 weeks of KD onset |
| 193 | d1_date_ucg6 | D | Date of ultrasonic cardiogram at 1 month of KD onset |
| 194 | d1_date_ucg2m | D | Date of ultrasonic cardiogram at 2 months of KD onset |
| 195 | d1_date_ucg7 | D | Date of ultrasonic cardiogram at 3 months of KD onset |
| 196 | d1_date_ucg8 | D | Date of ultrasonic cardiogram at 6 months of KD onset |
| 197 | d1_date_ucg9 | D | Date of ultrasonic cardiogram at 12 months of KD onset |
| 198 | d2_lmca0 | N | LMCA in ultrasonic cardiogram before IVIG administration |
| 199 | d2_lmca5 | N | LMCA in ultrasonic cardiogram at 2 weeks of KD onset |
| 200 | d2_lmca6 | N | LMCA in ultrasonic cardiogram at 1 month of KD onset |
| 201 | d2_lmca2m | N | LMCA in ultrasonic cardiogram at 2 months of KD onset |

| 202 | d2_lmca7 | N | LMCA in ultrasonic cardiogram at 3 |
|-----|----------|---|------------------------------------------|
| | | | months of KD onset |
| 203 | d2_lmca8 | N | LMCA in ultrasonic cardiogram at 6 |
| | | | months of KD onset |
| 204 | d2_lmca9 | N | LMCA in ultrasonic cardiogram at 12 |
| | | | months of KD onset |
| 205 | d3_lad0 | N | LAD in ultrasonic cardiogram before IVIG |
| | | | administration |
| 206 | d3_lad5 | N | LAD in ultrasonic cardiogram at 2 weeks |
| | | | of KD onset |
| 207 | d3_lad6 | N | LAD in ultrasonic cardiogram at 1 month |
| | | | of KD onset |
| 208 | d3_lad2m | N | LAD in ultrasonic cardiogram at 2 months |
| | | | of KD onset |
| 209 | d3_lad7 | N | LAD in ultrasonic cardiogram at 3 months |
| | | | of KD onset |
| 210 | d3_lad8 | N | LAD in ultrasonic cardiogram at 6 months |
| | | | of KD onset |
| 211 | d3_lad9 | N | LAD in ultrasonic cardiogram at 12 |
| | | | months of KD onset |
| 212 | d4_lcx0 | N | LCX in ultrasonic cardiogram before IVIG |
| | | | administration |
| 213 | d4_lcx5 | N | LCX in ultrasonic cardiogram at 2 weeks |
| | | | of KD onset |
| 214 | d4_lcx6 | N | LCX in ultrasonic cardiogram at 1 month |
| | | | of KD onset |
| 215 | d4_lcx2m | N | LCX in ultrasonic cardiogram at 2 months |
| | | | of KD onset |
| 216 | d4_lcx7 | N | LCX in ultrasonic cardiogram at 3 months |

| | | | of KD onset |
|-----|---------------|---|------------------------------------------|
| 217 | d4_lcx8 | N | LCX in ultrasonic cardiogram at 6 months |
| | | | of KD onset |
| 218 | d4_lcx9 | N | LCX in ultrasonic cardiogram at 12 |
| | | | months of KD onset |
| 219 | d5_rca_prox0 | N | Proximal segment of RCA in ultrasonic |
| | | | cardiogram before IVIG administration |
| 220 | d5_rca_prox5 | N | Proximal segment of RCA in ultrasonic |
| | | | cardiogram at 2 weeks of KD onset |
| 221 | d5_rca_prox6 | N | Proximal segment of RCA in ultrasonic |
| | | | cardiogram at 1 month of KD onset |
| 222 | d5_rca_prox2m | N | Proximal segment of RCA in ultrasonic |
| | | | cardiogram at 2 months of KD onset |
| 223 | d5_rca_prox7 | N | Proximal segment of RCA in ultrasonic |
| | | | cardiogram at 3 months of KD onset |
| 224 | d5_rca_prox8 | N | Proximal segment of RCA in ultrasonic |
| | | | cardiogram at 6 months of KD onset |
| 225 | d5_rca_prox9 | N | Proximal segment of RCA in ultrasonic |
| | | | cardiogram at 12 months of KD onset |
| 226 | d6_rca_mid0 | N | Middle segment of RCA in ultrasonic |
| | | | cardiogram before IVIG administration |
| 227 | d6_rca_mid5 | N | Middle segment of RCA in ultrasonic |
| | | | cardiogram at 2 weeks of KD onset |
| 228 | d6_rca_mid6 | N | Middle segment of RCA in ultrasonic |
| | | | cardiogram at 1 month of KD onset |
| 229 | d6_rca_mid2m | N | Middle segment of RCA in ultrasonic |
| | | | cardiogram at 2 months of KD onset |
| 230 | d6_rca_mid7 | N | Middle segment of RCA in ultrasonic |
| | | | cardiogram at 3 months of KD onset |

| 231 | d6_rca_mid8 | N | Middle segment of RCA in ultrasonic |
|-----|-----------------------|---|--------------------------------------------|
| | | | cardiogram at 6 months of KD onset |
| 232 | d6_rca_mid9 | N | Middle segment of RCA in ultrasonic |
| | | | cardiogram at 12 months of KD onset |
| 233 | el_ecg0 | С | ECG before IVIG administration |
| 234 | e1_ecg_txt0 | Т | Text of ECG before IVIG administration |
| 235 | el_ecg1 | С | ECG after IVIG administration |
| 236 | el_ecg_txtl | Т | Text of ECG after IVIG administration |
| 237 | e2_xray0 | С | X-ray before IVIG administration |
| 238 | e2_xray_txt0 | Т | Text of X-ray before IVIG administration |
| 239 | e2_xray1 | С | X-ray after IVIG administration |
| 240 | e2_xray_txt1 | Т | Text of X-ray after IVIG administration |
| 241 | e3_mra0 | С | MRA before IVIG administration |
| 242 | e3_mra_txt0 | Т | Text of MRA before IVIG administration |
| 243 | e3_mra1 | С | MRA after IVIG administration |
| 244 | e3_mra_txt1 | Т | Text of MRA after IVIG administration |
| 245 | e4_mpi0 | С | Myocardial perfusion imaging before IVIG |
| | | | administration |
| 246 | e4_mpi_txt0 | Т | Text of myocardial perfusion imaging |
| | | | before IVIG administration |
| 247 | e4_mpi1 | С | Myocardial perfusion imaging after IVIG |
| | | | administration |
| 248 | e4_mpi_txt1 | Т | Text of myocardial perfusion imaging after |
| | | | IVIG administration |
| 249 | ae | В | Adverse events |
| 250 | f1_infection | В | Serious infection |
| 251 | fl_infection_hour | N | Occurrence time of serious infection |
| 252 | fl_infection_duration | N | Duration of serious infection |
| 253 | fl_infection_relation | С | Relation between serious infection and |

| | | | drugs |
|---|---|---|---|
| 254 | fl_infection_intensity | С | Intensity of serious infection |
| 255 | fl_infection_treat | С | Treatment of serious infection |
| 256 | fl_infection_dose | N | Dose adjustment of serious infection |
| 257 | fl_infection_t1 | Т | Time to start the adjustment of serious |
| | | | infection |
| 258 | fl_infection_t2 | Т | Time to end the adjustment of serious |
| | | | infection |
| 259 | fl_infection_outcome | N | Outcome of serious infection |
| 260 | f2_skin | В | Skin allergy |
| 261 | f2_skin_hour | N | Occurrence time of skin allergy |
| 262 | f2_skin_duration | N | Duration of skin allergy |
| 263 | f2_skin_relation | С | Relation between skin allergy and drugs |
| 264 | f2_skin_intensity | С | Intensity of skin allergy |
| 265 | f2_skin_treat | С | Treatment of skin allergy |
| 266 | f2_skin_dose | N | Dose adjustment of skin allergy |
| 267 | f2_skin_t1 | D | Time to start the adjustment of skin allergy |
| 268 | f2_skin_t2 | D | Time to end the adjustment of skin allergy |
| 269 | f2_skin_outcome | С | Outcome of skin allergy |
| 270 | f3_heartfailure | В | Heart failure |
| 271 | f3_heartfailure_hour | N | Occurrence time of heart failure |
| 272 | f3_heartfailure_duration | N | Duration of heart failure |
| 273 | f3_heartfailure_relation | С | Relation between heart failure and drugs |
| 274 | f3_heartfailure_intensity | С | Intensity of heart failure |
| 275 | f3_heartfailure_treat | С | Treatment of heart failure |
| 276 | f3_heartfailure_dose | N | Dose adjustment of heart failure |
| 277 | f3_heartfailure_t1 | D | Time to start the adjustment of heart |
| | | | failure |
| 278 | f3_heartfailure_t2 | D | Time to end the adjustment of heart failure |

| 279 | f3_heartfailure_outcome | С | Outcome of heart failure |
|---|---|---|---|
| 280 | f4_thromb | В | Thrombogenesis |
| 281 | f4_thromb_hour | N | Occurrence time of thrombogenesis |
| 282 | f4_thromb_duration | N | Duration of thrombogenesis |
| 283 | f4_thromb_relation | С | Relation between thrombogenesis and |
| | | | drugs |
| 284 | f4_thromb_intensity | С | Intensity of thrombogenesis |
| 285 | f4_thromb_treat | С | Treatment of thrombogenesis |
| 286 | f4_thromb_dose | N | Dose adjustment of thrombogenesis |
| 287 | f4_thromb_t1 | D | Time to start the adjustment of |
| | | | thrombogenesis |
| 288 | f4_thromb_t2 | D | Time to end the adjustment of |
| | | | thrombogenesis |
| 289 | f4_thromb_outcome | С | Outcome of thrombogenesis |
| 290 | f5_hypertension | В | Hypertension |
| 291 | f5_hypertension_hour | N | Occurrence time of hypertension |
| 292 | f5_hypertension_duration | N | Duration of hypertension |
| 293 | f5_hypertension_relation | С | Relation between hypertension and drugs |
| 294 | f5_hypertension_intensity | С | Intensity of hypertension |
| 295 | f5_hypertension_treat | С | Treatment of hypertension |
| 296 | f5_hypertension_dose | N | Dose adjustment of hypertension |
| 297 | f5_hypertension_t1 | D | Time to start the adjustment of |
| | | | hypertension |
| 298 | f5_hypertension_t2 | D | Time to end the adjustment of |
| | | | hypertension |
| 299 | f5_hypertension_outcome | С | Outcome of hypertension |
| 300 | f6_othae | В | Other adverse events |
| 301 | f6_othae_txt | Т | Text of other adverse events |
| 302 | f6_othae_hour | N | Occurrence time of other adverse events |

| 303 | f6_othae_duration | N | Duration of other adverse events |
|-----|--------------------|---|-------------------------------------------|
| 304 | f6_othae_relation | С | Relation between other adverse events and |
| | | | drugs |
| 305 | f6_othae_intensity | С | Intensity of other adverse events |
| 306 | f6_othae_treat | С | Treatment of other adverse events |
| 307 | f6_othae_dose | N | Dose adjustment of other adverse events |
| 308 | f6_othae_t1 | D | Time to start the adjustment of other |
| | | | adverse events |
| 309 | f6_othae_t2 | D | Time to end the adjustment of other |
| | | | adverse events |
| 310 | f6_othae_outcome | С | Outcome of other adverse events |
| 311 | f7_death | В | Death due to adverse events |
| 312 | f7_death_time | N | Occurrence time of death due to adverse |
| | | | events |
| 313 | ae_solve | В | Adverse events are solved or not |
| 314 | remedy | В | Remedy is used or not |
| 315 | remedy_ivig | В | Second IVIG administration in the remedy |
| 316 | remedy_ivig_dose | Т | Dose of second IVIG administration in the |
| | | | remedy |
| 317 | remedy_mp | В | Methylprednisolone in the remedy |
| 318 | remedy_mp_dose | Т | Dose of methylprednisolone in the remedy |
| 319 | remedy_ifx | В | Infliximab in the remedy |
| 320 | remedy_ifx_dose | Т | Dose of infliximab in the remedy |
| 321 | remedy_ims | В | Other immunosuppressants in the remedy |
| 322 | remedy_ims_dose | Т | Dose of other immunosuppressants in the |
| | | | remedy |
| 323 | remedy_pte | В | Plasma exchange in the remedy |
| 324 | remedy_oth | В | Other remedy |
| 325 | remedy_oth_txt | Т | Text of other remedy |

| 326 | date_tempcover | D | Date of final body temperature recovery |
|-----|-----------------|---|-----------------------------------------|
| 327 | date_revisit | D | Date of last revisit |
| 328 | compliance | В | Completing the protocol or not |
| 329 | quit_person | С | Proposer of quitting |
| 330 | quit_person_oth | Т | Other proposer of quitting |
| 331 | quit_reason | С | Reason of quitting |
| 332 | quit_reason_txt | Т | Text of other reason of quitting |
| 333 | date_crf | D | Date of CRF |

### 8. Reference

- 1. Dallaire F, Dahdah N. New Equations and a Critical Appraisal of Coronary Artery Z Scores in Healthy Children. J Am Soc Echocardiogr.2011;24(1):60 60-74.
- 2. McCrindle BW, Rowley AH, Newburger JW, et al. Diagnosis, Treatment, and Long-Term Management of Kawasaki Disease: A Scientific Statement for Health Professionals From the American Heart Association. Circulation 2017;135:e927-e99.
- 3. ZHU B H, LV H T, SUN L, et al. A meta-analysis on the effect of corticosteroid therapy in Kawasaki disease [J]. Eur J Pediatr, 2012, 171(3): 571-8.
- 4. Research Committee on Kawasaki Disease. Report of subcommittee on standardization of diagnostic criteria and reporting of coronary artery lesions in Kawasaki disease. Tokyo, Japan: Ministry of Health and Welfare, 1984. (In Japanese.)
- 5. Wang D, Pocock S. A win ratio approach to comparing continuous non-normal outcomes in clinical trials. Pharm Stat. 2016; 15:238-45.